CLINICAL TRIAL: NCT07388875
Title: A Single-arm, Phase II Study of Sacituzumab Tirumotecan Combined With Anlotinib in Patients With Extensive-stage Small Cell Lung Cancer After Failure of PD-(L)1 Inhibitor Plus Chemotherapy
Brief Title: Sacituzumab Tirumotecan Plus Anlotinib in Previously Treated ES-SCLC
Acronym: SKB264-ANLO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Xiujuan Qu, Professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOG2601
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Participants will receive sacituzumab tirumotecan in combination with anlotinib. Sacituzumab tirumotecan will be administered intravenously, and anlotinib will be administered orally, according to the dosing schedule specified in the study protocol. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined discontinuation criteria are met.
  Interventions: Drug: Sacituzumab Tirumotecan; Drug: Anlotinib

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan — Sacituzumab tirumotecan is an antibody-drug conjugate targeting Trop-2. It will be administered intravenously according to the dosing schedule specified in the study protocol. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined discontinuation criteria are met.
Drug: Anlotinib — Anlotinib is an oral small-molecule multi-target tyrosine kinase inhibitor. It will be administered orally according to the dosing regimen specified in the study protocol. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined discontinuation criteria are met.

SUMMARY:
This is a Phase II, single-arm, open-label clinical study to evaluate the efficacy and safety of Sacituzumab Tirumotecan (SKB264) combined with Anlotinib in patients with extensive-stage small cell lung cancer (ES-SCLC). The study is designed for patients who have experienced disease progression or treatment failure after prior first-line therapy with a PD-(L)1 inhibitor combined with platinum-based doublet chemotherapy. The primary hypothesis is that this combination therapy will improve the objective response rate compared to historical controls.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is an aggressive malignancy with a poor prognosis. While chemotherapy combined with immunotherapy is the standard first-line treatment for extensive-stage SCLC (ES-SCLC), therapeutic options remain limited for patients who progress after this initial therapy. There is an urgent need to explore new treatment strategies to extend patient survival.

Sacituzumab Tirumotecan (SKB264) is a humanized antibody-drug conjugate (ADC) targeting TROP2, which is often overexpressed in SCLC. It works by delivering a topoisomerase I inhibitor directly to tumor cells. Anlotinib is a multi-target tyrosine kinase inhibitor that suppresses tumor angiogenesis and proliferation.

This study investigates the potential synergistic effect of combining SKB264 with Anlotinib. The rationale is that anti-angiogenic therapy (Anlotinib) may normalize tumor vasculature, thereby enhancing the delivery and efficacy of the ADC (SKB264) within the tumor microenvironment.

Eligible participants will receive Sacituzumab Tirumotecan (200 mg intravenously on Day 1 of each 3-week cycle) combined with Anlotinib (8 mg orally once daily on Days 1-14 of each 3-week cycle). The study utilizes a Simon's two-stage minimax design to assess the Objective Response Rate (ORR) as the primary endpoint. Secondary objectives include evaluating Progression-Free Survival (PFS), Overall Survival (OS), and the safety profile of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing informed consent; male or female.
* Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC).
* Disease progression after receiving only one prior line of therapy consisting of a PD-(L)1 inhibitor combined with platinum-based doublet chemotherapy.
* At least one measurable target lesion per RECIST v1.1 as assessed by the investigator, which has not been previously irradiated.
* Patients with asymptomatic brain metastases, or patients with treated brain metastases and stable symptoms for ≥4 weeks, are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ and bone marrow function (no blood transfusion, recombinant human thrombopoietin, or colony-stimulating factors within 2 weeks prior to first dose), defined as follows:
* Hematologic function:
* Absolute neutrophil count ≥1.5 × 10⁹/L
* Platelet count ≥100 × 10⁹/L
* Hemoglobin ≥90 g/L
* Hepatic function:
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN; for patients with liver metastases, AST and ALT ≤5 × ULN
* Albumin ≥30 g/L
* Total bilirubin ≤1.5 × ULN
* Renal function:
* Creatinine clearance ≥50 mL/min, calculated using the Cockcroft-Gault formula
* Coagulation function:
* International normalized ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) ≤1.5 × ULN
* Women of childbearing potential and men with partners of childbearing potential must agree to use effective medical contraception from signing informed consent until 6 months after the last dose of study treatment.
* Subjects must voluntarily participate in the study, provide written informed consent, and be able to comply with protocol-required visits and study procedures.

Exclusion Criteria:

* Participation in another interventional drug clinical trial within 4 weeks prior to enrollment.
* Tumors with a high risk of massive hemoptysis, as judged by the investigator.
* Prior systemic anti-tumor therapy with anti-angiogenic agents.
* Prior treatment with TROP2-targeted therapies and/or topoisomerase I inhibitors.
* History of other malignancies within the past 5 years, except for adequately treated cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
* Known hypersensitivity or allergy to any investigational product or its components.
* Known positive human immunodeficiency virus (HIV) infection, history of acquired immunodeficiency syndrome (AIDS), or known active syphilis infection.
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Receipt of live vaccines within 30 days prior to the first dose of study treatment.
* History of interstitial lung disease (ILD) or non-infectious pneumonitis requiring steroid treatment; current ILD or non-infectious pneumonitis; or suspected ILD or non-infectious pneumonitis that cannot be excluded by imaging at screening. Severe pulmonary impairment due to pulmonary comorbidities, including but not limited to:
* Pulmonary embolism within 3 months prior to first dose
* Severe asthma
* Severe chronic obstructive pulmonary disease
* Restrictive lung disease
* Pleural effusion
* Autoimmune, connective tissue, or inflammatory diseases involving the lungs (e.g., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis)
* Prior pneumonectomy
* Active autoimmune disease requiring systemic treatment within the past 2 years (hormone replacement therapy is not considered systemic treatment, such as type 1 diabetes mellitus, hypothyroidism requiring only thyroid hormone replacement, or adrenal or pituitary insufficiency requiring physiologic doses of corticosteroids).
* Active infection requiring systemic therapy within 2 weeks prior to the first dose of study treatment.
* Serious concomitant diseases that, in the investigator's judgment, may compromise patient safety or interfere with completion of the study, including but not limited to uncontrolled hypertension, severe diabetes mellitus, or active infection.
* Documented severe dry eye syndrome, severe meibomian gland dysfunction and/or blepharitis, or a history of corneal disorders that may interfere with delayed corneal healing.
* Pregnant or breastfeeding women; women of childbearing potential with a positive baseline pregnancy test; or women of childbearing potential who are unwilling to use effective contraception during study treatment and for 6 months after the last dose of study treatment.
* Any other condition that, in the investigator's opinion, makes the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the first dose of study treatment until disease progression, intolerance, or start of new anti-cancer therapy, assessed every 6 weeks for the first 12 months and every 12 weeks thereafter, up to approximately 24 months.
  Objective response rate (ORR) as assessed by the investigator according to RECIST version 1.1, defined as the proportion of patients achieving complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the first dose of study treatment until disease progression, intolerance, or start of new anti-cancer therapy, assessed every 6 weeks for the first 12 months and every 12 weeks thereafter, up to approximately 24 months
  The time from the first dose of study treatment to the first documented disease progression or death from any cause.
Overall Survival (OS) | From first dose until death, assessed every 6 weeks (Year 1) then every 12 weeks, and every 3 months during survival follow-up, up to approximately 24 months.
  The time from randomization (or first dose) to death from any cause.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is ongoing and the data are considered confidential. Data sharing may be considered after study completion upon reasonable request and approval by the sponsor.